CLINICAL TRIAL: NCT01304433
Title: Evaluation on the Safety Profile of Hydroxyethyl Starch (HES) 130/0.42
Brief Title: Safety Profile of Hydroxyethyl Starch
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HC-O-H-0811
Record Dates: First submitted 2011-02-21; First posted 2011-02-25 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Plasma Volume Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: hydroxyethyl starch (HES) 130/0.42
  Interventions: Drug: Venofundin 6% / Tetraspan 6%

INTERVENTIONS:
Drug: Venofundin 6% / Tetraspan 6% — Venofundin 6% / Tetraspan 6%

SUMMARY:
The study is primarily aimed to collect further data on the safety of the investigational product in a large patient population when used in routine clinical practice in the Asian-Pacific region.

ELIGIBILITY:
Inclusion:

* patients with ASA risk score ≤ III,
* non-emergency patients, i.e. elective surgery

Exclusion:

* contraindications as listed for HES 130/0.42

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
number of adverse drug reactions | up to 48 hours

SECONDARY OUTCOMES:
change in haemodynamics during surgery or intensive care unit stay | up to 48 hours

CONTACTS AND LOCATIONS:
Locations (6):
- China (5):
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu Province
  - The Sixth Hospital of Shanghai, Shanghai
  - The First Hospital of Shanghai, Shanghai
  - Dong Fang Gan Dan Hospital of Shanghai, Shanghai
- Hospital Kuala Lumpur, Kuala Lumpur, Malaysia, Malaysia